CLINICAL TRIAL: NCT01227876
Title: Assessment of Clinical Efficacy of 1% Prednisolone Acetate (Ster ®), Produced by união química, Compared to 1% Prednisolone Acetate (Pred ® Fort), Produced by Allergan, in the Control of Postoperative Inflammation in Cataract Surgery.
Brief Title: Clinical Efficacy of the Drug Ster® Compared With Predfort® in Control of Postoperative Inflammation in Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREUNI0710; Version 01
Record Dates: First submitted 2010-10-15; First posted 2010-10-25 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Inflammation; Cataract Surgery
Keywords: PREUNI0710; cataract
MeSH Terms: conditions — Inflammation; Cataract | interventions — Triclosan; Methylprednisolone

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Test (Experimental): Ster ® (prednisolone 1% ophthalmic suspension - União Química)
  Interventions: Drug: Ster
- Comparator (Active Comparator): Pred Fort ® (prednisolone 1% ophthalmic suspension - Allergan)
  Interventions: Drug: Pred Fort

INTERVENTIONS:
Drug: Ster — prednisolone 1% ophthalmic suspension
  Arms: Test
Drug: Pred Fort — prednisolone 1% ophthalmic suspension
  Arms: Comparator

SUMMARY:
Is the primary objective of this investigation to compare the clinical efficacy of the drug test - Ster ® (prednisolone 1% ophthalmic suspension - Union Chemicals) in the comparator - Fort ® Pred (prednisolone 1% ophthalmic suspension - Allergan) in the control of postoperative inflammation in cataract surgery by phacoemulsification through periodic measurement of efficiency scores (number of cells in the anterior chamber, the presence of fibrin in the anterior chamber, conjunctival hyperemia, corneal edema and Descemet folds).

DETAILED DESCRIPTION:
The secondary objective is to compare the safety data observed during the study period, ie will be assessed the frequency and intensity of adverse reactions and compared statistically between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree with all study procedures and sign, by his own free will, IC;

  * Adult patients, regardless of gender, ethnicity or social status, with good mental health;
  * Patients who present at screening visit, a clinical diagnosis of cataract with an indication for corrective surgery with phacoemulsification technique.

Exclusion Criteria:

* Patients with a history or clinical diagnosis of other eye diseases such as glaucoma, corneal ulcers, scarring, and uveitis;

  * Patients with known hypersensitivity to any component of the drug under investigation;
  * Patients who have made use of systemic corticosteroids within 15 days before surgery;
  * Patients who have made use of topical corticosteroids in the 7 days before surgery;
  * Patients who have made use of systemic antibiotics in the 15 days preceding surgery;
  * Patients who have made use of topical antibiotics in the 7 days before surgery;
  * Patients presenting abnormality, at the discretion of the principal investigator in the following ophthalmic examinations Preoperative slit-lamp examination, measurement of intraocular pressure (applanation tonometry) and examination of background, other than the underlying disease (cataract);
  * Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Comparison of clinical efficacy between the test and comparator drugs by measuring periodic scores of efficacy in established clinical parameters. | 28 days of treatment.
  We will evaluate the clinical parameters of number of cells in the anterior chamber, the presence of fibrin in the anterior chamber, conjunctival hyperemia, corneal edema and Descemet folds.The treatment will last for 28 days following the conduct of routine postoperative cataract. There will be a total of 04 returns after surgery and with them 07, 14, 21 and 28 days. On each return, will register the change of parameters of efficacy and safety.

SECONDARY OUTCOMES:
Comparison of safety data observed during the study period by assessing frequency and intensity of adverse reactions, compared statistically between groups. | 28 days of treatment.
  The treatment will last for 28 days following the conduct of routine postoperative cataract. There will be a total of 04 returns after surgery and with them 07, 14, 21 and 28 days. On each return, will register the change of parameters of efficacy and safety.

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil